CLINICAL TRIAL: NCT04635904
Title: Imagery Based Interventions for the Treatment of Anxiety Related Disorders: Mechanisms and Optimizing Outcomes
Brief Title: Imagery Rescripting and Imaginal Exposure for Social Anxiety: Mechanisms and Outcomes in an Analog Sample
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Jonathan D. Huppert, Professor, PhD, Certified Clinical Psychologist, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: isf2157/2020
Record Dates: First submitted 2020-11-08; First posted 2020-11-19 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Social Anxiety
Keywords: Social anxiety symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor that assess mental imagery content (see secondary outcomes) are blind to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaginal exposure (Experimental): A behavioral intervention in imagery
  Interventions: Behavioral: Imaginal exposure one-session
- Imagery rescripting (Experimental): A different behavioral intervention in imagery
  Interventions: Behavioral: Imagery rescriptinf one-session

INTERVENTIONS:
Behavioral: Imaginal exposure one-session — Participants in this arm will be asked to decide alongside with the intervention provider (a clinical PhD student or M.A student under the supervision of the principal investigator) to imagine a script based on a future distressing anxiety provoking scenarios multiple times while honing in on the most negative aspects.
  Arms: Imaginal exposure
Behavioral: Imagery rescriptinf one-session — Participants in this arm will be asked to decide alongside with the intervention provider (a clinical PhD student or M.A student under the supervision of the principal investigator) o imagine a script based on a future distressing anxiety provoking scenarios one time while honing in on the most negative aspects. Afterwards they will insert changes into the script that try to help them cope in the imagery.
  Arms: Imagery rescripting

SUMMARY:
This study will recruit 100 participants who self-report high symptoms of social anxiety (Social phobia inventory >30). Participants will be randomly assigned to receive either one analog intervention of Imagery Rescripting (IR) or Imaginal Exposure. We will test the efficacy and mechanisms behind each interventions.

DETAILED DESCRIPTION:
After being informed about the study potential risks, all patients giving written informed consent will undergo screening to determine eligibility for study entry. They will be randomly assigned to two conditions (Imagery rescripting Vs. Imaginal exposure) at a 1:1 ratio. Participants will attend three ~1 hour online ZOOM sessions (pre-assessment and measurement, intervention, and post assessment and measurement).

Assessors will be blind to the treatment condition.

ELIGIBILITY:
Inclusion Criteria: SPIN scores >= 30 -

Exclusion Criteria:

can't report a negative imagery related to a future social scenario. Attending active psychotherapy sessions.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Social phobia inventory (SPIN) at the follow-up session | Will be measured at Baseline (6,9, or 12 days before intervention), Post-intervention (immediately after the intervention) and Follow-up ( 7 days after the intervention)
  The SPIN is a validated self-report instrument assessing average social phobia symptom intensity over the past week. possible scores range from 0 (not at all) to 4 (Extremly).
  change = (follow-up score - Baseline Score)

SECONDARY OUTCOMES:
Change from Baseline in the Thought fusion inventory (TFI) at the follow-up session | Will be measured at Baseline (6,9, or 12 days before intervention), Post-intervention (immediately after the intervention) and Follow-up ( 7 days after the intervention)
  The TFI is a validated 14 item self-reported instrument assessing average belief in statement that describe the effects of thoughts on reality, objects and actions. Possible scores range from 0 (Do not believe at all) to 100 (completely convinced it is true) in intervals of 10.
  change = Follow-up - Baseline Score.
Change from Baseline in the White Bear Suppresion inventory (WBSI) at the follow-up session | Will be measured at Baseline (6,9, or 12 days before intervention), Post-intervention (immediately after the intervention) and Follow-up ( 7 days after the intervention)
  The WBSI is a validated 15 item self-reported instrument assessing average tendency to suppress mental thoughts. Possible scores range from 0 (Do not agree) to 5 (very much agree).
  change = Follow-up - Baseline Score.
Change from Baseline in the Positive and Negative Affect Scale (PANAS) international version short form (10 items from the negative subscale only) at the follow-up session | Will be measured at Baseline (6,9, or 12 days before intervention) and Follow-up ( 7 days after the intervention)
  The PANAS International short form is a validated 10 item self-reported instrument assessing emotions after at a certain point in time. Possible scores range from 0 (Not at all) to 5 (Extremely). It will be assessed right after the participant describes the script.
  change = Follow-up - Baseline Score.
Change from Baseline to follow-up in the amount of negative and positive/neutral content details the participant provides while describing the negative imagery. The imagery will be probed using the Waterloo Image and Memories Interview (WIMI). | Will be measured at Baseline (6,9, or 12 days before intervention) and Follow-up ( 7 days after the intervention)
  The WIMI is a validated 10 item interview for assessing content of imagery. valence of the details will be scored using a trained coder. change = Follow-up - Baseline Score.
Change from Baseline to follow-up in negativity of the core-beliefs that the participant link to the negative imagery provided in the WIMI. | Will be measured at Baseline (6,9, or 12 days before intervention) and Follow-up ( 7 days after the intervention)
  The WIMI is a validated 10 item interview for assessing content of imagery and core-beliefs.
  Core beliefs are related to the participant perception of himself, others and the world.
  valence of the beliefs will be scored using a trained coder. change = Follow-up - Baseline Score.
imaginal Behavioral Approach Test (iBAT) that measures the participant's willingness to interact with pre-scripted distressing scenarios in imagination | Will be measured at Baseline (6,9, or 12 days before intervention) and Follow-up ( 7 days after the intervention)
  The iBAT is currently being developed in our lab. The more levels the participants passes (listen to imaginal scenario in full without pressing "skip") the higher the score (from 0 to 10)
  Recruitment is under way and pre-registration is available at the open science frame work website:
  https://osf.io/bp42h/?view_only=5211617cedf94f71a4daa746e98d924a
Sentence Completion Task (SCT). Measures participants automatic interpretation bias while being presented with 10 ambiguous social scenarios. | Will be measured at Baseline (6,9, or 12 days before intervention) and Follow-up ( 7 days after the intervention)
  The SCT has been found to correlate with social anxiety symptoms and differentiate between clinical and non clinical population.
  participants enters words that complete scenario described in a sentence. Participant's answers are coded to negative, positive and neutral valence. Then, the participant ratio negative bias is calculated from 0 (complete positive bias) to 1 (complete negative bias)
The Patient's Experience of Attunement and Responsiveness Scale (PEAR) measures participants' feelings of acceptance by the intervention and interview providers | Will be measured at Baseline (6,9, or 12 days before intervention), Post-intervention (immediately after the intervention) and Follow-up ( 7 days after the intervention)
  the PEAR is a well validated self-report instrument. It has 20 items total. Each item is scored from 0 (not at all) to 3 (very much)
The Brief core schema scale (BCSS) measures participants' self beliefs about themselves and others. | Will be measured at Baseline (6,9, or 12 days before intervention), Post-intervention (immediately after the intervention) and Follow-up ( 7 days after the intervention)
  the BCSS is a well validated self-report instrument. It has 24 items total. Each item is scored from 1 (believe it slightly) to 3 (believe it totally)
Change across time in the Mini Social phobia inventory - revised (mini SPIN-R) from baseline to pre-treatment and from pre-treatment to follow-up. | Daily, from Baseline to follow-up (a total of 14, 17, or 20 days)
  The Mini SPIN-R is a validated self-report instrument assessing average social phobia symptom intensity over the past day. possible scores range from 0 (not at all) to 4 (Extremly).
  measured once at the end of each day.
Daily questionnaire about negative intrusive imagery in general and specific to the imagery provided in the interview. | Daily, from Baseline to follow-up (a total of 14, 17, or 20 days)
  Participants are asked alongside the MINI-SPIN-R (see above) whether they had negative imagery during that day (In general) or the specific image they provided (specific). If the report they did experience images they rate two items from the TFI and two items from WBSI adapted for daily measurment. One item about feelings of mastery on the image. 4 items from the BCSS (2 related to the self, one negative and one positive and 2 related to others, one negative and one positive belief). With regards to the specific image they also report on a 0-100 analog scale how vivid, intrusive, distressing that image was for them.

OTHER OUTCOMES:
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) | Baseline only
  This interview is based on DSM-5 diagnostic criteria. It will allow us to detect the presence of social anxiety disorder before the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Huppert, PhD, Principal Investigator — Professor
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aderka IM, Pollack MH, Simon NM, Smits JA, Van Ameringen M, Stein MB, Hofmann SG. Development of a brief version of the Social Phobia Inventory using item response theory: the Mini-SPIN-R. Behav Ther. 2013 Dec;44(4):651-61. doi: 10.1016/j.beth.2013.04.011. Epub 2013 May 3. PMID 24094790
- [Background] Connor KM, Davidson JR, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). New self-rating scale. Br J Psychiatry. 2000 Apr;176:379-86. doi: 10.1192/bjp.176.4.379. PMID 10827888
- [Background] Muris P, Merckelbach H, Horselenberg R. Individual differences in thought suppression. The White Bear Suppression Inventory: factor structure, reliability, validity and correlates. Behav Res Ther. 1996 May-Jun;34(5-6):501-13. doi: 10.1016/0005-7967(96)00005-8. PMID 8687372
- [Background] Romano M, Moscovitch DA, Saini P, Huppert JD. The effects of positive interpretation bias on cognitive reappraisal and social performance: Implications for social anxiety disorder. Behav Res Ther. 2020 Aug;131:103651. doi: 10.1016/j.brat.2020.103651. Epub 2020 May 22. PMID 32504886
- [Background] Moscovitch DA, Vidovic V, Lenton-Brym AP, Dupasquier JR, Barber KC, Hudd T, Zabara N, Romano M. Autobiographical memory retrieval and appraisal in social anxiety disorder. Behav Res Ther. 2018 Aug;107:106-116. doi: 10.1016/j.brat.2018.06.008. Epub 2018 Jun 22. PMID 29960125
- [Background] Tolin DF, Gilliam C, Wootton BM, Bowe W, Bragdon LB, Davis E, Hannan SE, Steinman SA, Worden B, Hallion LS. Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders. Assessment. 2018 Jan;25(1):3-13. doi: 10.1177/1073191116638410. Epub 2016 Mar 17. PMID 26988404